CLINICAL TRIAL: NCT02156271
Title: Mechanisms of Sleep Latency and Health: The Effect of a Melatonin Receptor Agonist in Inflammation and Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00013501
Record Dates: First submitted 2014-05-30; First posted 2014-06-05 (Estimated); Results first posted 2014-12-09 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2014-05

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ramelteon (Active Comparator): Subjects will take ramelteon 8mg one time daily 30 minutes before bedtime with approximately 8 ounces of water. Subjects have a 2 out of 3 chance of receiving ramelteon.
  Interventions: Drug: ramelteon
- placebo (Placebo Comparator): 15 subjects will be randomized to receive the placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ramelteon
  Other Names: Rozerem
  Arms: ramelteon
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to help scientist better understand the effect of a 12-week single daily evening dose of ramelteon (Rozerem ©), a drug that has been approved by the U. S. Food and Drug Administration (FDA) for the treatment of insomnia (trouble falling asleep or staying asleep). The study will measure levels of inflammation, fasting insulin and fasting glucose (sugar) in subjects who are taking either ramelteon (8 mg) or placebo.

ELIGIBILITY:
Inclusion Criteria:

At screening visit:

* aged 18-65
* nonsmokers
* for women: oral contraceptive (OC) or hormone replacement therapy (HRT) nonusers

To schedule the baseline PSG (Visit 2), subjects must meet the following inclusion criteria:

* ages 18-65 inclusive;
* PSQI-Component 2 (sleep latency) score of greater than 1;
* non-smoker (e.g., less than 20 cigarettes in the past 5 years);
* habitual bedtime between 8:30 pm and midnight
* For premenopausal women:

  * regular menstrual cycles determined by Framingham Study criteria;
  * not pregnant and no history of oral contraceptive (OC) usage in last 6-months.
* For postmenopausal women:

  * no recent (< 6 months) use of Hormone Replacement Therapy (HRT)
  * no surgical menopause

Exclusion Criteria:

* positive urine drug screen
* Potential subjects with hypersensitivity to ramelteon or any components of the formulation will be excluded from participation.
* Given that ramelteon should not be used by individuals with severe hepatic impairment, or in patients in combination with fluvoxamine, individuals who report liver problem or use of fluvox will be excluded.
* use of rifampin (Rifadin ©); ketoconazole (Nizora ©l); or fluconazole (Diflucan ©).
* Ramelteon has not been studied in children or adolescents, and the effects in these populations are unknown, thus only individuals above 18 years will participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 75 subjects signed consent and were enrolled in the study. Of these, 23 (31%) failed to qualify to participate in the study based on screening assessments, 12 (16%) withdrew consent prior to randomization, and 4 (5%) dropped out before randomization. As a result, 39 subjects were randomized.
Groups:
- Ramelteon: Subjects will take ramelteon 8mg one time daily 30 minutes before bedtime with approximately 8 ounces of water. Subjects have a 2 out of 3 chance of receiving ramelteon.
  ramelteon
- Placebo: 15 subjects will be randomized to receive the placebo
  placebo
Period: Overall Study
Arm/Group | Ramelteon | Placebo
Started | 26 | 13
Completed | 22 | 10
Not Completed | 4 | 3
Not completed — Physician Decision | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon | Placebo | Total
Number analyzed (Participants) | 26 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 13 | 39
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 26 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Sleep Onset Latency (SOL) as Measured by Self Report (Sleep Diary)
Description: The average of a week of sleep onset latency data from the sleep diary filled out in the morning by the participating subjects. Sleep latency is defined as the length of time it takes from lying down for the night until sleep onset.
Time Frame: Day 89-90
Measure: Least Squares Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 22 | 10
minutes | 29.7 (21.7) | 24.8 (15.2)

2. Primary Outcome: Mean Latency to Persistent Sleep (LPS) Via Polysomnography
Description: Elapsed time from the beginning of the Polysomnography recording to the onset of the first 20 minutes of continuous sleep was measured.
Time Frame: Day 89-90
Measure: Least Squares Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 22 | 10
minutes | 19.2 (11.3) | 48.6 (33.0)

3. Primary Outcome: Change in Metabolic Syndrome (MetSyn)
Time Frame: Baseline, Day 30, Day 60, Day 89-90
Population: Data was not collected, and therefore not analyzed.
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Sleep Onset Latency (SOL) as Measured by Pittsburgh Sleep Qualtiy Index (PSQI)
Description: Subjects completed component 2 of the PSQI questionnaire. Component 2 asks questions about sleep latency and is scored on a scale from 0 (better) to 3 (worse).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 26 | 13
units on a scale | 2.5 (0.7) | 2.8 (0.6)

5. Secondary Outcome: Change in Total Sleep Time
Description: Change in sleep time will be determined by PSG.
Time Frame: Day -1-0, Day 89-90
Population: Data was not collected, and therefore not analyzed.
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Inflammatory Biomarkers C-reactive Protein (CRP)
Time Frame: Day 89-90
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 22 | 10
ng/mL | 11.9 (12.7) | 7.3 (28.1)

7. Secondary Outcome: Interleukin 6 (IL-6)
Time Frame: Day 89-90
Measure: Least Squares Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 22 | 10
pg/mL | 2.2 (1.4) | 1.3 (1.0)

8. Secondary Outcome: Insulin Resistance (IR)
Description: In each subject, an insulin resistance score based on Homeostasis Model Assessment (HOMA-IR) was estimated at day 89-90. Formula: fasting plasma glucose (mmol/l) times fasting serum insulin (mU/l) divided by 22.5. Low HOMA-IR values indicate high insulin sensitivity, whereas high HOMA-IR values indicate low insulin sensitivity (insulin resistance).
Time Frame: Day 89-90
Measure: Least Squares Mean (Standard Deviation); unit: HOMA-IR value
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 22 | 10
HOMA-IR value | 12.6 (12.2) | 7.9 (6.6)

9. Primary Outcome: Sleep Onset Latency (SOL) as Measured by Pittsburgh Sleep Qualtiy Index (PSQI)
Description: as for outcome 4
Time Frame: day 89 - 90
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 22 | 10
units on a scale | 1.72 (0.9) | 0.93 (1.1)

10. Primary Outcome: Mean Latency to Persistent Sleep (LPS) Via Polysomnography
Description: as for outcome 2
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 26 | 13
minutes | 41.0 (25.4) | 46.3 (20.1)

11. Primary Outcome: Sleep Onset Latency (SOL) as Measured by Self Report (Sleep Diary)
Description: The average of a week of sleep onset latency data from the sleep diary filled out in the morning by the participating subjects.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 26 | 13
minutes | 41.3 (32.9) | 38.8 (19.8)

12. Secondary Outcome: Inflammatory Biomarkers C-reactive Protein (CRP)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 26 | 13
mg/L | 11.8 (16.9) | 26.1 (38.9)

13. Secondary Outcome: Insulin Resistance (IR)
Description: In each subject, an insulin resistance score based on Homeostasis Model Assessment (HOMA-IR) was estimated at baseline. Formula: fasting plasma glucose (mmol/l) times fasting serum insulin (mU/l) divided by 22.5. Low HOMA-IR values indicate high insulin sensitivity, whereas high HOMA-IR values indicate low insulin sensitivity (insulin resistance).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: HOMA-IR value
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 26 | 13
HOMA-IR value | 16.9 (10.8) | 12.4 (9.2)

14. Secondary Outcome: Interleukin 6 (IL-6)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 26 | 13
pg/mL | 1.6 (1.1) | 2.5 (2.4)

ADVERSE EVENTS:
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/13
Other Adverse Events (participants affected / at risk) | 8/26 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramelteon (N=26) | Placebo (N=13)
Dizziness (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Body Aches (General disorders) | 0 | 1
Drowsiness (Nervous system disorders) | 4 | 0
Back Ache (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Sore Ankle (Musculoskeletal and connective tissue disorders) | 1 | 0
cold symptoms (General disorders) | 1 | 0
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
dislocated shoulder (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes